CLINICAL TRIAL: NCT03976388
Title: Virtual Clinical Simulation Amongst Undergraduate Medical Students
Brief Title: Virtual Clinical Simulation for Training Amongst Undergraduate Medical Students: A Pilot Randomised Trial
Acronym: VIRTUE-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: Hospital de Simulación, Universidad Andres Bello (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez Lomakin, Principal Investigator, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UNAB-001
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Medical Education
Keywords: Virtual reality; Clinical simulation; Adherence; Guidelines

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors, analysts and investigators will be masked in this trial. Due to the intervention's characteristics, it has been deemed impossible to mask participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical virtual simulator (Experimental): A clinical virtual simulator contains an interactive medical case depicting an acutely ill patient seeking care at the emergency department. The case will be delivered in small groups (up to 6 participants) in sessions lasting up to 20 minutes. After the simulation has been completed, a feedback session lasting up to 30 minutes will be delivered as well.
  Interventions: Device: Clinical Virtual Simulator
- Standard educational session (Active Comparator): A small-group discussion (up to 6 participants) using patients with the same condition as the one selected for the clinical simulator will be held for participants allocated to the control group. These sessions will be led by a physician and have a maximum duration of up to 60 minutes.
  Interventions: Other: Small-Group Discussion

INTERVENTIONS:
Device: Clinical Virtual Simulator — Interactive medical case delivered using touch-sensitive screens in small group sessions.
  Other Names: BodyInteract(R)
  Arms: Clinical virtual simulator
Other: Small-Group Discussion — Small group discussion led by a physician.
  Arms: Standard educational session

SUMMARY:
In this trial, undergraduate medical students will be randomised to undergo training using a virtual reality simulator (BodyInteract®) or a standard small-group interactive discussion of a clinical scenario. Adherence to current clinical recommendations will be considered as primary outcomes for this study.

DETAILED DESCRIPTION:
Objective: To assess whether a virtual reality simulator might facilitate learning and improve adherence to current clinical guidelines. Methodology: A double-masked randomised trial will be held among students at the School of Medicine of the Universidad Andres Bello. Participants will be randomised to receive training using a clinical virtual simulator (Body Interact®, Body Interact Inc, Austin, TX) designed to review key concepts in Cardiology. Students allocated to the control group will receive a small-group discussion lasting up to 60 minutes in which key topics regarding the same clinical condition will be reviewed as well. Main outcomes include the overall performance in an objective structured clinical examination (OSCE) that will be reviewed by an expert panel prior to its implementation and adherence to specific recommendations in current national guidelines. This OSCE will be held 15 days after the educational session has taken place. Analyses will be undertaken under the intention to treat principle and missing data will be handled using multiple imputation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical student at the Universidad Andrés Bello
* Currently undergoing the 4th or 5th year of medical training in Chile
* Obtained a passing grade in Cardiology for general physicians.

Exclusion Criteria:

* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with passing grades in an Objective Structured Clinical Examination (OSCE) | 2 weeks after attending the educational session.
  Number of participants with marks over 60% in an OSCE.
Marks attained in an Objective Structured Clinical Examination (OSCE) | 2 weeks after attending the educational session.
  Marks attained in an OSCE depicting the clinical scenario described in educational sessions. In this examination, the implementation of diagnostic and therapeutic interventions will score marks that will then be compared between groups.
Adherence to guideline recommendations | 2 weeks after attending the educational session.
  Adherence to specific recommendations in national guidelines relevant to the diagnosis and management of the clinical condition being studied.

SECONDARY OUTCOMES:
Time to solve the clinical scenario | 2 weeks after attending the educational session.
  Time required to solve the clinical scenario depicted in the Objective Structured Clinical Examination
Time to deliver specific interventions | 2 weeks after attending the educational session.
  Time required to implement specific diagnostic and therapeutic interventions relevant to the clinical scenario

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Martinez, MD, MSc, Study Director — Universidad Andres Bello
Locations (1):
- Hospital de Simulación, Universidad Andrés Bello, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook DA, Hatala R, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hamstra SJ. Technology-enhanced simulation for health professions education: a systematic review and meta-analysis. JAMA. 2011 Sep 7;306(9):978-88. doi: 10.1001/jama.2011.1234. PMID 21900138
- [Background] Lopreiato JO, Sawyer T. Simulation-based medical education in pediatrics. Acad Pediatr. 2015 Mar-Apr;15(2):134-42. doi: 10.1016/j.acap.2014.10.010. PMID 25748973
- [Background] Li L, Yu F, Shi D, Shi J, Tian Z, Yang J, Wang X, Jiang Q. Application of virtual reality technology in clinical medicine. Am J Transl Res. 2017 Sep 15;9(9):3867-3880. eCollection 2017. PMID 28979666
- [Background] Edvardsen O, Steensrud T. [Virtual reality in medical education]. Tidsskr Nor Laegeforen. 1998 Feb 28;118(6):902-6. Norwegian. PMID 9543805